CLINICAL TRIAL: NCT03663569
Title: Changes in Clinical Control of COPD Patients Measured by the Clinical COPD Questionnaire During Therapy With Spiolto®Respimat® in Routine Clinical Practice
Brief Title: A Study on the Control of Chronic Obstructive Pulmonary Disease (COPD) in Patients Taking the Combination of Tiotropium and Olodaterol Using the Respimat® Inhaler
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1237-0072
Record Dates: First submitted 2018-07-26; First posted 2018-09-10 (Actual); Results first posted 2020-10-22 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- subjects with COPD
  Interventions: Drug: Spiolto® Respimat®

INTERVENTIONS:
Drug: Spiolto® Respimat® — Drug

SUMMARY:
Open-label observational study which includes COPD patients that are receiving treatment with Spiolto® Respimat® for approximately 6 weeks, which is the average time between two medical consultations.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to participation
* Female and male patients ≥40 years of age
* Patients diagnosed with COPD and based upon the investigator's decision requiring a new prescription of Spiolto Respimat® (combination of two long-acting bronchodilators) according to Spiolto® Respimat® SmPC, GOLD COPD Strategy Document 2018 (GOLD COPD groups B to D) and local COPD guidelines

Exclusion Criteria:

* Patients with contraindications according to Spiolto® Respimat® SmPC
* Patients already on a LABA/LAMA combination (free and fixed dose) in the last 6 weeks before study entry
* Patients continuing LABA/ICS treatment should not be additionally treated with Spiolto® Respimat® in order to avoid a double dosing of long-acting beta-agonists
* Pregnancy and lactation
* Current participation in any clinical trial or any other non-interventional study of a drug or device.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Around 4500 COPD patients from approximately 11 countries will be collected, with a signed informed consent will be maintained in the ISF at the investigational site irrespective of whether they have been treated or not.
Sampling Method: Non-Probability Sample
Enrollment: 4819 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2019-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Medvedchikov, +431801057896, Study Chair — alexey.medvedchikov@boehringer-ingelheim.com
Locations (388):
- Bulgaria (17):
  - MBAL Sveti Ivan Rilski-2003, Dupnitsa
  - SBALBB "Pencho Semov" - Gabrovo EOOD, Gabrovo
  - SBALPFZ Haskovo EOOD, Haskovo
  - MBAL Kiro Popov EOOD, Karlovo
  - MBAL Sv. Ivan Rilski EOOD, Kozloduy
  - MBAL "Prof. Dr P. Stoyanov" AD - Mihail Kirov, Lovech
  - Iliana Valkanova, Plovdiv
  - MBAL Sveti Panteleimon, Plovdiv
  - "Medical Center-Razgrad"OOD, Razgrad
  - Medical Center Re Spiro OOD, Razgrad
  - MBAL Sliven to VMA Sofia, Sliven
  - Grigor Lalov, Smolyan
  - SBALPFZ-Sofia district EOOD, Sofia
  - Prevencia 2000 MCDMP OOD, Stara Zagora
  - Medical Center "Research expert" OOD, Varna
  - Medical Center "Tara" OOD, Veliko Tarnovo
  - MC"Sv.Ivan Rilski"OOD, Vidin
- Czechia (77):
  - MUDr. Alena Jelinkova, Bílina
  - MUDr. Eva Krizova, Boskovice
  - Ambulance pro nemoci plicni a TBC, s.r.o., Brno
  - Jana Jančíková, Brno
  - MUDr Hana Vašínová, Brno
  - MUDr. Ilona Binkova, Brno
  - MUDr. Jana Slapnickova s.r.o., Brno
  - MUDr. Jaroslava Lovakova, Brno
  - MUDr. Michal Svarc, Broumov
  - MUDr. Martin Polasek, CeskyTesinKonakov
  - Plicní Čáslav s.r.o., Čáslav
  - MUDr. Jan Faktor Medipont s.r.o., České Budějovice
  - MUDr. Josef Hlavac Medipont s.r.o., České Budějovice
  - MUDr. Renata Bilkova, Děčín
  - MUDr. Jiri Guthwirth, Dobřís
  - MUDr. Martin Adamec Alergonet Group, Frýdek-Místek
  - MUDr. Marie Buresova, Havlíčkův Brod
  - MUDr. Jana Psikalova, Holešov
  - MUDr. Stanislava Bednarova, Holešov
  - MUDr. Petr Šafránek, Hořovice
  - MUDr. Hana Lochmanova AXIMED s.r.o., Hradec Králové
  - MUDr. Ales Bohac Plicni ambulance, Hranice
  - MUDr. Lenka Fousova, Hustopece U Brna
  - MUDr. Bohumil Kralicek, Jihlava
  - MUDr. Jirina Knillova, Jihlava
  - MUDr. Alexandra Woznicova, Jirkov
  - MUDr. Michaela Baerova, Kosmonosy
  - MUDr. Petr Kolman, Kyjov
  - MUDr. Milanda Sipkova, Liberec
  - Plucni Ambulance Louny s.r.o., Louny
  - MUDr. Ilona Pavlisova, s.r.o., Miroslav
  - MUDr. Michaela Baerova, Mlada Boreslav
  - MUDr. Pavla Shihatova, Náchod
  - MUDr. Dusan Velart, Nový Jičín
  - MUDr. Sarka Hofrova, Nový Jičín
  - MUDr. Sarka Klimesova, Nymburk
  - MUDr. Ondrej Sobotik, Olomouc
  - MUDr. RAdoslav Alexa, Orlová - Lutyně
  - MUDr. Milena Sramkova, Ostrava
  - MUDr. Jana Balounova, Ostrava
  - MUDr. Jana Kocianova, Ostrava
  - Plicní-ambulance Terezie Janásková, s.r.o, Ostrava, Bělský Les
  - MUDr. Tereza Dobesova Aximed s.r.o., Pardubice
  - MUDr. Miluse Zitkova, Pardubice
  - MUDr. Jiri Zoula Aries Medici s.r.o., Pelhřimov
  - MUDr. Petr Hartman, Pilsen
  - MUDr. Jitka Smolova, Pilsen
  - MUDr. Vladimir Makrlik, Pilsen
  - MUDr. Petr Šafránek, Pilsen
  - MUDr. Andrea Svabkova, Pilsen
  - MUDr. Jana Janková Zátopková, Poděbrady
  - MUDr. Olga Krizova, Pohořelice
  - První plicní ambulance s.r.o., Prague
  - MUDr. Fransitek Petrik, Prague
  - MUDr. Romana Davidova, Prague
  - MUDr. Iva Stachova, Prague
  - MUDr. Ivana Zatloukalova, Prague
  - MUDr. Milada Typltová, Prague
  - MUDr. Ivana Jirmanova, Prague
  - MUDr. Jana Jirouskova, Prague
  - MUDr. Lenka Povysilova, Prague
  - MUDr. Vera Reichmanova, Prague
  - MUDr. Vera Pacovska, Prague
  - MUDr. Bronislava Viest, Prague
  - MUDr. Ivana Boučková, Prague
  - MUDr. Romana Ivankova, Prostějov
  - MUDr. Helena Ringlerova, Rokycany
  - MUDr. Jaroslav Mares, Strakonice
  - MUDr. Margit Hóracková, Šumperk
  - MUDr. Alena Kortusova, Ústí nad Labem
  - MUDr. Olga Martinkovicova, Ústí nad Labem
  - MUDr. Pavel Stach, Valašské Meziříčí
  - MUDr. Eva Sabova, Veselí nad Moravou
  - MUDr. Pavel Matuska, Zábřeh
  - MUDr. Jiri Dolecek, Žamberk
  - MUDr. Michal Pasler, Žamberk
  - MUDr. Alena Prochazkova, Židlochovice
- Hungary (35):
  - Ecce Homo Orvosi Bt., Balassagyarmat
  - Dr. Major Katalin IZOPULM Kft., Budapest
  - FOKUSZ-PULMO Egeszsegügyi, Kutatasi, Oktatoi Tanacsado Bt, Budapest
  - Kineto-Med Bt., Budapest
  - Dr. Szabó Gyöngyi, Budapest
  - Dr. Szilvia Vasas, Budapest
  - Emósi Bt., Budapest
  - Főv.XIX.ker.Önk.Egészségügyi Int, Budapest
  - Dr. Zoltan Gyula Bende, Budapest
  - Fenykepzeles KFT, Csitár
  - Electro-Medic Bt., Debrecen
  - Rizikó '99, Debrecen
  - Szent Pantaleon Hospital, Dunaújváros
  - Pulmo Bt., Edelény
  - Dr. Gyetvainé Dr. Lanczki Éva, Eger
  - Dr. Kontz Katalin, Gyöngyössolymos
  - Dr. Szász Zoltán, Győr
  - Györ Tüdögondozo, Győr
  - Broncho-Vin BT., Gyula
  - Pulmoport Kft., Gyula
  - Rakvács-Mózes Bt., Kaposvár
  - Selye János Kórház, Rendelőintézet, Tüdőgondozó, Komárom
  - Sz.-Sz.-B. MK és EOK. Mátészalka, Mátészalka
  - Borsod-Abaúj-Zemplén Megyei Központ Kórház és Egyetemi Oktatókórház Semmelweis Tagkórház, Miskolc
  - Dr. Bíró Margit, Monok
  - Monor Szakrendelö Tüdögondozo, Monor
  - Infer-Med Kft, Nagykozár
  - Dr. Varga Ágnes, Pécs
  - Ujpesti Szakorvosi Rendelöintezet, Pócsmegyer
  - Dr. Anna Bartha, Siófok
  - Dr. Breining és Társa Egészségügyi Szolgáltató Bt., Sopron
  - Dr. Radeczky Éva, Százhalombatta
  - Dr. Bánvölgyi Aranka Milassinné, Szeged
  - Dr. Geherne Dr. Huszar Hermina Eveline, Szombathely
  - Szabolcs-Szatmár-Bereg Megyei Kórházak és Egyetemi Oktatókórház, Vásárosnamény
- Israel (23):
  - ASSUTA Ashdod Ltd., Ashdod
  - Barzilai Medical Center, Ashkelon
  - Clalit - Bat Yam, Bat Yam
  - Soroka Medical Center, Beersheba
  - Hillel Yaffe Medical Center, Hadera
  - Carmel Medical Center, Haifa
  - Edith Wolfson Medical Center, Holon
  - Maccabi Healthcare, Holon
  - Shaarei Zedek Medical Center, Jerusalem
  - Research Fund of the Hadassah Medical Organization (R.A.), Jerusalem
  - Clalit - Jerusalem East, Jerusalem East
  - Meir Medical Center Israel, Kfar Saba
  - Holy Family Hospital, Nazareth
  - Rabin Medical Center (Beilinson Hospital), Petah Tikva
  - Clalit Health Services, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Health Corporation of the Ziv Medical Center (R.A.), Safed
  - Clalit - Nazareth, Tel Aviv
  - Clalit - Rishon, Tel Aviv
  - Clalit - Carmiel, Tel Aviv
  - Sheba Medical Center, Tel-Hashomer / Ramat Gan
  - PORIYA Medical Center, Tiberias
  - Assaf Harofeh MC, Zrifin
- Lithuania (5):
  - Hospital of Lithuanian University of Health Sciences Kauno klinikos, Kaunas
  - Klaipeda Hospital, Klaipėda
  - Enterprise Klaipeda University Hospital, Klaipėda
  - Vilnius University Hospital Santaros klinikos, Vilnius
  - Public Enterprise Vilnius District Central Outpatient Clinic, Vilnius
- Poland (48):
  - ISPL Beata Kuklińska, Bialystok
  - Specjalistyczy Gabinet Lekarski Urszula Świetlik Malesa, Biała Podlaska
  - Poradnia Chorób Płuc Samodzielny Publiczny Zakład Opieki Zdrowotnej"Szpital Powiatowy"W Bochni, Bochnia
  - Indywidualna Praktyka Lekarska Aleksandra Burysz, Bydgoszcz
  - Specjalistyczna Praktyka Lekarska Choroby Płuc Agata Kalicka, Bydgoszcz
  - Indywidualna Specjalistyczna Praktyka Lekarska Dr. n. med. Szymon Dworniczak, Chorzów
  - Indywidualna Specjalistyczna Praktyka Lekarska Anna Góra-Florek, Ciecierzyn
  - ODM Gdynia, Gdynia
  - Gabinet lekarski Renata Pejas-Dulewicz, Gmina Końskie
  - Specjalistyczna Praktyka Lekarska i USG, Jasło
  - Specjalistyczny Gabinet Lekarski Juliusz Bokiej, Jelenia Góra
  - Niepubliczny Zakład Opieki Specjalistycznej "Zdrowe Płuca", Kielce
  - Indywidualna Specjalistyczna Praktyka Lekarska lek. Krzysztof Lis, Kielce
  - Specjalistyczny Zespół Gruźlicy i chorób Płuc, Koszalin
  - Gabinet lekarski Wojciech Machowiak, Kościan
  - Poradnia Chorób płuc, Krakow
  - Indywidualna Praktyka Lekarska Aleksander Kania, Krakow
  - Gabinet lekarski Thomasz Mysior, Krakow
  - Lekarskie Wizyty Domowe Jarosław Zięba, Kłomnice
  - Uniwersytecki Szpital Kliniczny Nr 1, Lodz
  - Centrum Leczenia Chorób Płuc w Łodzi, Lodz
  - Przychodnia Specjalistyczna Snzoz Med Med. Sp.Z O.O, Lodz
  - Specjalistyczna Praktyka Lekarska Piotr Kamiński, Lublin
  - Alergopneuma sp. Z.o.o., Lublin
  - ISPL Łukasz Minarowski, Olmonty
  - Prywatny gabinet lakarski Izabela Piętowska-Łazuka, Parczew
  - Medycyna-diagnostyka Adam Nowiński, Piaseczno
  - MEDICAL-MED. Indywidualna Specjalistyczna Praktyka Lekarska Barbara Kuźnar-Kamińska, Poznan
  - Indywidualna Specjalistyczna Praktyka Lekarska Magdalena Kostrzewska, Poznan
  - Poradnia Gruźlicy i Chorób Płuc SPZOZ Proszowice, Proszowice
  - Gabinet lekarski Roman Masarczyk, Pyskowice
  - Gabinet lekarski Edyta Kozińska, Płock
  - Szpital Rejonowy im.dr Rostka-Oddził Pulmonologiczny, Racibórz
  - Podkarpackie Centrum Chorób Płuc, Rzeszów
  - Gabinet lekarski Choroby płuc i oskrzeli Joanna Tęsiorowska, Sieradz
  - Indywidualna Specjalistyczna Praktyka Lekarska Krzysztof Filipek, Sosnowiec
  - NZOZ Poradnia Chorób Płuc i Alergologii, Słupsk
  - NZOZ Centrum Medyczne SBB, Tarnobrzeg
  - Viltis Medica Spejalistyczan Praktyla Lekarska lek.med. Agata Kot, Trzebnica
  - STANMED Gabinet Lekarski Robert Staniszewski, Warsaw
  - Instytut Gruźlicy i Chorób Płuc, Warsaw
  - Gabinet lekarski Beata Żołnowska, Warsaw
  - MSWiA, Warsaw
  - Wizyty Domowe Internisty B. Homola-Piekarska, Warsaw
  - Gabinet lekarski Andrzej Jaworski, Warsaw
  - Gabinet Internistyczny-Choroby płuc lek.med.M.Kraszewska, Wieruszów
  - Specjalistyczna Praktyka Lekarska dr n.med. Andrzej Obojski, Wroclaw
  - Specjalistyczny Szpital Chorób Płuc Odrodzenie im Klary Jelskiej, Zakopane
- Romania (28):
  - DaniPneumoMed SRL, Arad
  - Butacel F. Maria Danisia - Medic Specialist Pneumolog, Bacau
  - Manolache Cristina - Medic Specialist Pneumologie, Bistrița
  - Dr. Bendas Magdalena, Botoșani
  - Muresan Alina Pneumoconsult Srl, Brasov
  - Dr Cosei Valentin-Caius Pfi, Bucharest
  - Borcea Corina-Ioana Persoana Fizica Autorizata, Bucharest
  - Ispas Elena-Irina Medic Specialist Pneumolog, Bucharest
  - Pneumo Clinic Care SRL, Constanța
  - Crm Pneumology Srl, Craiova
  - Nicolosu Med Srl, Craiova
  - Avencord SRL, Focşani
  - Miron V. Ramona - Medic Colaborator, Iași
  - Howas Med Srl, Jud Constanta
  - Ciumarnean G Lorena Medic Specialist, Jud. Cluj, Mun. Cluj-Napoca
  - Chis P Ana Florica - Medic Specialist Pneumologie, Jud. Cluj, Mun. Cluj-Napoca
  - Cabinet Medical Individual Defta I. Doina-Elisabeta, Jud. Giurgiu , Mun. Giurgiu
  - Rarcolmed Srl, Milcovul
  - Vlad M. Elena - Medic Primar Pneumolog, Mun. Târgu Jiu
  - Medic Primar Pneumologie Stoleru Manuela, Piatra Neamţ
  - Raissa Maria Medical Srl, Popeşti-Leordeni
  - PFI Chirea C. Monica Valentina, Râmnicu Sărat
  - Viosan-Resp S.R.L., Râmnicu Vâlcea
  - Jager Pneumo Services Srl, Sat Ariniș
  - Sc Nexus Medical Srl, Sat Visan, Jud Iasi
  - Cabinet Medical Individual Dr. Butuc Lilia, Tg.Lăpuș
  - Cabinet Medical Pneumologie Dr. Albu Claudia, Timișoara
  - CMI Dr. Mihailescu Constantin, Vânju-Mare
- Russia (122):
  - Treatment and consultation center, Angarsk
  - Volga district hospital, Astrakhan
  - Alexander Mariinsky regional clinical hospital, Astrakhan
  - Departmental clinical hospital on the station Barnaul of OJSC "RZhD", Barnaul
  - Barnaul city hospital Nr.5, Barnaul
  - Out-patient hospital "Harmony of health", Belgorod
  - Bryansk regional hospital No. 1, Bryansk
  - Chekhov central district out-patient hospital, Checkov 2
  - Chelyabinsk regional clinical hospital, Chelyabinsk
  - Road clinical hospital at station Chelyabinsk RRR, Chelyabinsk
  - LLC "AllergoStop", Center of asthma prophylactic and treatment of allergy and asthma, Chelyabinsk
  - Regional Clinical Hospital Nr.3, Chelyabinsk
  - Institution of public health City clinical hospital #11, Chelyabinsk
  - Regional oncology dispensary, Irkutsk
  - Irkutsk state clinical hospital Nr.1, Irkutsk
  - East and Siberian institute of medical and ecological studies, Irkutsk
  - LLC Pulsar, Iskitim
  - City clinical hospital No. 4, Ivanovo
  - Kaluga regional clinical hospital, Kaluga
  - LLC "City Clinical hospital #12", Kazan'
  - Medical Association "Spasenie", Kazan'
  - City clinical hospital Nr. 16, Kazan'
  - State autonomy institution of public health, Kazan'
  - Kemerovo regional clinical phthisiopulmonology medical center, Kemerovo
  - Regional clinical hospital of emergency medical care named after M.A. Podgorbunsky, Kemerovo
  - LLC "Doctor Lite", Kirov
  - Kirov clinical and diagnostic centeron the basis of out-patient hospital Nr. 1, Kirov
  - Krai clinical hospital Nr. 1 named after prof. S.V. Ochapovskogo, Krasnodar
  - Krai clinical hospital, Krasnoyarsk
  - Krasnoyarsk inter-district clinical hospital Nr. 20 named after I.S. Berzon, Krasnoyarsk
  - Kurgan out-patient hospital, Kurgan
  - Kurgan regional clinical hospital, Kurgan
  - Out-patient hospital of regional budgetary institution of public health, Kursk
  - Medassist-K, Kursk
  - Lipetsk city out-patient hospital Nr. 7, Lipetsk
  - Republican clinical hospital of war and labor veterans, Makhachkala
  - Educational institution of higher education named after N.I. Pirogov of Ministry of health of Russia, Moscow
  - Moscow scientific and clinical educational center for respiratory medicine, Moscow
  - City out-patient hospital Nr. 22 of department of public health of Moscow, branch Nr. 2, Moscow
  - City out-patient hospital Nr. 134 of department of public health of Moscow, Moscow
  - City out-patient hospital Nr. 52 of department of public health of Moscow, Moscow
  - First Moscow State Medical University named after I. M. Sechenov, Moscow
  - Institution of public health "City out-patient hospital #180 of department of public health of Moscow, Moscow
  - Consultation and diagnostic center Nr. 6 of department of public health of Moscow, Moscow
  - Moscow Regional Research Clinical Institute named after M.F. Vladimirsky, Moscow
  - Nizhnevartovsk county hospital No.2, Nizhnevartovsk
  - Nizhny Novgorod scientific and research institute of sanitary science and occupational pathology, Nizhny Novgorod
  - Privolzhsky Research Medical University, Nizhny Novgorod
  - Nizhny Novgorod city clinical hospital named after N.A. Semashko, Nizhny Novgorod
  - Novokuznetsk city clinical hospital Nr. 29, Novokuznetsk
  - Azbuka zdoroviya, Novosibirsk
  - Road clinical hospital on station Novosibirsk-Main of OJSC "RZhD", Novosibirsk
  - City clinical hospital No. 2, Novosibirsk
  - Zdorovaya Semiya, Novosibirsk
  - Scientific and research institute of physiology and fundamental medicine, Novosibirsk
  - City clinical out-patient hospital No. 1, Novovsibirsk
  - Clinical medical sanitary station Nr. 7, Omsk
  - City out-patient hospital No. 2, Omsk
  - Multifunctional center of modern medicine "Evromed", Omsk
  - ZAO "Multifunctional center of modern medicine "Evromed", Omsk
  - Orenburg regional clinical hospital No. 2, Orenburg
  - City hospital named after S. P. Botkin, Oryol
  - Penza regional clinical hospital named after N.N. Burdenko, Penza
  - Clinical hospital No. 6 named after G.A. Zakhariyn, Penza
  - City clinical out-patient hospital of Perm, Perm
  - Perm clinical center of federal medical and biological agency "Medical sanitary station #140" on the basis of out-patient hospital #2, Perm
  - City clinical out-patient hospital #2, Perm
  - "City out-patient hospital #7" on the basis of out-patient hospital #2, Perm
  - City clinical out-patient hospital No. 4, Perm
  - Perm regional clinical hospital, Perm
  - Hospital of Karelia republic named after V.A.Baranov, Petrozavodsk
  - 1586 military clinical hospital of Ministri of Public Defense, Podolsk
  - Treatment and prophylactic institution of union health resort "Rodnik", Pyatigorsk
  - Clinical and diagnostic center "Zdorovie" of Rostov-on-Don, Rostov-on-Don
  - Rostov regional clinical hospital, Rostov-on-Don
  - City clinical hospital No. 20 of Rostov-on-Don", Rostov-on-Don
  - Regional clinical cardiology dispensary, Ryazan
  - Regional clinical hospital, Ryazan
  - ZAO "Medi", Saint Petersburg
  - LLC "Medical center XXI century" Bryanseva 13", Saint Petersburg
  - Aleksandrovskaya City Hospitel, Saint Petersburg
  - City Consultative and Diagnostic Centre Nr. 1, Saint Petersburg
  - Institute of Medical Trials, Saint Petersburg
  - First Saint-Petersburg state medical university named after acad. I.P.Pavlov, Saint Petersburg
  - Samara city out-patient hospital No.1, Samara
  - Samara medical and sanitary unit Nr. 5 of the Kirovsky district, Samara
  - City clinical hospital Nr 4 of Samara, Samara
  - Samara city hospital Nr. 13 of Zheleznodorozhny district, Samara
  - Samara city clinical out-patient hospital No.15, Samara
  - National Mordovia research state university named after N.P. Ogarev, Saransk
  - Saratov city out-patient hospital Nr. 9, Saratov
  - Saratov city clinical hospital No. 8, Saratov
  - Saratov city out-patient hospital Nr. 10, Saratov
  - Simferopol city clinical hospital Nr. 7, Simferopol
  - Simferopol clinical hospital, Simferopol
  - Out-patient hospital #5, Smolensk
  - Clinical hospital No. 1, Smolensk
  - Stavropol krai clinical hospital, Stavropol
  - Tambov regional clinical hospital named after V.D. Babenko, Tambov
  - Tolyatti city hospital Nr. 5, Tolyatti
  - Treatment and diagnostic center, Tomsk
  - Out-patient hospital No. 1, Tomsk
  - Tomsk Regional clinical hospital, Tomsk
  - Federal state budgetary institution of SibFNKC FMBA of Russia, Tomsk
  - City hospital Nr. 9, Tula
  - Regional Clinical Hospital, Tver'
  - Regional hospital No. 19 Out-patient hospital, Tyumen
  - City clinical hospital Nr. 21, Ufa
  - Republican clinical hospital named after G.G. Kuvatov, Ufa
  - Vladimir Regional clinical hospital, Vladimir
  - Volgograd regional clinical hospital Nr. 1, Volgograd
  - Non-state institution of public health Divisional clinical hospital on station Volgograd-1 of OJSC "RZhD", Volgograd
  - Institution of public health of Voronezh region "Voronezh regional clinical consultation and diagnostic center", Voronezh
  - LLC medical center "Diagnostic plus", Voronezh
  - Institution of public health of Yaroslavl region Regional clinical hospital, Yaroslavl
  - LLC Medical unity "Novaya Bolnitsa, Yekaterinburg
  - Sverdlovsk regional hospital Nr. 2, Yekaterinburg
  - Central city clinical hospital No. 1 of Oktyabrsky district, Yekaterinburg
  - City clinical hospital No. 14, Yekaterinburg
  - Central clinical hospital Nr. 3, Yekaterinburg
  - Medical Association "Novaya Bolnitsa" Polyclinic, Yekaterinburg
  - Central City Hospital Nr.7, Yekaterinburg
- Slovenia (19):
  - Internistična ambulanta za pljučne in alergijske bolezni Karmen Kramer Vrščaj, Celje
  - Pulmološka ambulanta dr. Snežana Ulčar Kostič s.p., Kamnik
  - MEDICOINTERNA, medicinske storitve in svetovanje, d.o.o., Kočevje
  - VELOG, Zdravstveni center, d.o.o., Kranj
  - Zdravstvene storitve in svetovanje, Tjaša Šubic s.p., Kranj
  - Verboten Kopriva Renata - Ordinacija Interne Medicine, Litija
  - Arjana Maček d.o.o, Ljubljana
  - Kambič-Kafol d.o.o., Ljubljana
  - Medvital Katarina Vukelič s.p., Ljubljana
  - Alveola, internistični ambulantni diagnostični center d.o.o., Maribor
  - CIIM PLUS, center za interno in interventno medicino, d.o.o., Maribor
  - INTERNIST MB - specialistična ambulantna dejavnost, Marko Bombek s.p., Maribor
  - Zdravstveno svetovanje in storitve, Krstić Zoran, s.p., Maribor
  - Mag. Anton Lopert, dr.med. - Zasebna internistična ambulanta, Murska Sobota
  - Zasebna ambulanta za pljučne bolezni, mag. Alojz Horvat, dr. med., Murska Sobota
  - Prim. mag. Šegota Nikša, dr.med., specialistična zdravniška dejavnost, s.p., Škofja vas
  - Dr. Ana Novakovic, Velenje
  - Dr. med. Tomaz Smonkar, Velenje
  - Dr. Mikro Lekic, Velenje
- Switzerland (7):
  - Gruppenpraxis Basel, Basel
  - Gruppenpraxis Frick, Frick
  - Gruppenpraxis Emmenbrücke, Geuensee
  - Berner Reha Zentrum Medizin Pneumologie, Heiligenschwendi
  - Gruppenpraxis Luzern, Lucerne
  - Spital Linth, Utznach
  - Zürcher RehaZentrum Wald, Wald
- Ukraine (7):
  - Dnipropetrovsk 6 City clinical Hospital, Dnipropetrovsk
  - Regional centre of Phtysiology and Pulmonology, Ivano-Frankivsk
  - City Clinical Hospital Nr. 13, Kharkiv
  - National Institute of Phthisiology and Pulmonology named F. G. Yanovsky National Academy of Medical Sciences of Ukraine, Kyiv
  - Volyn Regional Clinical Hospital, Lutsk
  - Lviv Regional Phthisiopneumological Clinical Treatment and Diagnostic Center, Lviv
  - Vinnytsia City Clinical Hospital Nr. 1, Vinnitsa

IPD SHARING:
Plan to Share IPD: Undecided
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions: 1. studiesin products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).Requestors can use the following link http://trials.boehringer-ingelheim.com/ to:
  1. find information in order to request access to clinical study data, for listed studies.
  2. request access to clinical study documents that meet criteria, and upon a signed 'Document Sharing Agreement'

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This open-label self-controlled observational study over an observational period of 6 weeks (2 visits) was to investigate the potential changes in clinical control of Chronic Obstructive Pulmonary Disease (COPD) patients measured by the Clinical COPD Questionnaire (CCQ) during treatment with Spiolto® Respimat® in routine practice.
Pre-assignment Details: All patients were screened for eligibility prior to participation in the trial. Patients attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
Groups:
- Spiolto® Respimat®: Chronic Obstructive Pulmonary Disease (COPD) patients administered a fixed dose combination of tiotropium and olodaterol (2.5 micrograms and 2.5 micrograms per puff) through Spiolto® Respimat® according to Spiolto® Respimat® Summary of Product Characteristics (SmPC) and the Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines for 6 weeks.
Period: Overall Study
Arm/Group | Spiolto® Respimat®
Started | 4819
Completed | 4756
Not Completed | 63
Not completed — Discontinuation of study | 11
Not completed — Never taken Spiolto® Respimat® | 1
Not completed — Deceased patient | 6
Not completed — Lost to Follow-up | 18
Not completed — Withdrawal of consent | 5
Not completed — Patient's request | 11
Not completed — Adverse Event | 4
Not completed — Not come to second visit | 3
Not completed — Not meet inclusion / exclusion criterion | 3
Not completed — Serious adverse event | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS): All screened patients with informed consent, date of registration (date of creation of screening form in the Electronic Case Report Form (eCRF)), and at least one documented administration of Spiolto® Respimat®.
Arm/Group | Spiolto® Respimat®
Number analyzed (Participants) | 4819
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.38 (9.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1459
  Male | 3360
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Therapeutic Success of Spiolto® Respimat® Treatment at Visit 2
Description: Therapeutic success of Spiolto® Respimat® treatment was defined as 0.4 point decrease in the Clinical Chronic Obstructive Pulmonary Disease (COPD) Questionnaire - Clinical COPD Questionnaire (CCQ) score from visit 1 to visit 2. Each of the 10 CCQ questions is scored by the patient on a 7-point scale between 0 (Never/Not limited at all) and 6 (Almost all the time/Totally limited or unable to do) at baseline (Visit 1) and at the end of the observation after approximately 6 weeks (Visit 2). The sum of the scores divided by 10 gives the CCQ score, which measures the health and functional status. A higher CCQ score is indicative of worse status.
Time Frame: At Visit 2 (6 weeks after baseline visit 1)
Population: Full analysis set (FAS): All screened patients with informed consent, date of registration (date of creation of screening form in the Electronic Case Report Form (eCRF)), at least one documented administration of Spiolto® Respimat®, and available total CCQ score at visit 1 and visit 2.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Spiolto® Respimat®
Number analyzed (Participants) | 4700
Percentage of participants | 81.38 [80.24 to 82.49]

2. Secondary Outcome: Changes in the Clinical COPD Questionnaire (CCQ) and the CCQ Symptom, Mental State and Functional State Domain Scores From Visit 1 (Baseline) to Visit 2
Description: The CCQ questionnaire contained 10 questions about symptoms, functional status and mental status. Each of the 10 CCQ questions was scored by the patient on a 7-point scale between 0 and 6 at baseline and at the end of observation after approximately 6 weeks. Symptom domain covered 4 questions (number 1, 2, 5, 6), Functional state domain covered 4 questions (number 7, 8, 9, 10), and Mental state domain covered 2 questions (number 3, 4). Scores for the questions in each domain were summed up and divided by the number of questions in each domain giving the resulting score for respective domain. The sum of the scores divided by 10 gives the CCQ score which measures the health and functional status. A higher CCQ score is indicative of worse status. Change of the score was calculated as visit 2 minus visit 1.
Time Frame: At baseline visit 1 and 6 weeks thereafter at visit 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Spiolto® Respimat®
Number analyzed (Participants) | 4700
Score on a scale
  Symptom | 1.09 (0.97)
  Functional state | 0.94 (0.96)
  Mental state | 1.04 (1.21)
  Total CCQ score | 1.02 (0.87)

3. Secondary Outcome: Physician's Global Evaluation (PGE) Score at Visit 1(Baseline)
Description: PGE score assessed the general condition of the patient on an 8-point ordinal scale from 1 (very poor) to 8 (excellent).
Time Frame: At visit 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Spiolto® Respimat®
Number analyzed (Participants) | 4700
Participants
  PGE score = 1 | 44
  PGE score = 2 | 471
  PGE score = 3 | 1176
  PGE score = 4 | 1428
  PGE score = 5 | 888
  PGE score = 6 | 539
  PGE score = 7 | 140
  PGE score = 8 | 14

4. Secondary Outcome: Physician's Global Evaluation (PGE) Score at Visit 2
Description: PGE score assessed the general condition of the patient on an 8-point ordinal scale from 1 (very poor) to 8 (excellent).
Time Frame: At visit 2 (6 weeks after baseline visit 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Spiolto® Respimat®
Number analyzed (Participants) | 4700
Participants
  PGE score = 1 | 3
  PGE score = 2 | 45
  PGE score = 3 | 212
  PGE score = 4 | 661
  PGE score = 5 | 1227
  PGE score = 6 | 1468
  PGE score = 7 | 891
  PGE score = 8 | 192
  Missing | 1

5. Secondary Outcome: Patient Overall Satisfaction With Spiolto® Respimat® Treatment at Visit 2
Description: Patient overall satisfaction with Spiolto® Respimat® treatment at visit 2 was reported.
Time Frame: At visit 2 (6 weeks after baseline visit 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Spiolto® Respimat®
Number analyzed (Participants) | 4700
Participants
  Very satisfied | 1474
  Satisfied | 2055
  Rather satisfied | 803
  Neither satisfied nor dissatisfied | 236
  Rather dissatisfied | 64
  Dissatisfied | 44
  Very dissatisfied | 20
  Not answered | 4

6. Secondary Outcome: Patient Satisfaction With Inhaling From the Respimat® Device at Visit 2
Description: Patient satisfaction with inhaling from the Respimat® device at visit 2 was reported
Time Frame: At visit 2 (6 weeks after baseline visit 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Spiolto® Respimat®
Number analyzed (Participants) | 4700
Participants
  Very satisfied | 1579
  Satisfied | 2119
  Rather satisfied | 694
  Neither satisfied nor dissatisfied | 211
  Rather dissatisfied | 49
  Dissatisfied | 30
  Very dissatisfied | 10
  Not answered | 8

7. Secondary Outcome: Patient Satisfaction With Handling of the Respimat® Inhalation Device at Visit 2
Description: Patient satisfaction with handling of the Respimat® inhalation device at visit 2 was reported.
Time Frame: At visit 2 (6 weeks after baseline visit 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Spiolto® Respimat®
Number analyzed (Participants) | 4700
Participants
  Very satisfied | 1554
  Satisfied | 2083
  Rather satisfied | 711
  Neither satisfied nor dissatisfied | 244
  Rather dissatisfied | 60
  Dissatisfied | 31
  Very dissatisfied | 11
  Not answered | 6

8. Secondary Outcome: Number of Participants Willing to Continue Treatment With Spiolto® Respimat® at Visit 2
Description: Number of participants willing to continue treatment with Spiolto® Respimat® at visit 2 was reported.
Time Frame: At visit 2 (6 weeks after baseline visit 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Spiolto® Respimat®
Number analyzed (Participants) | 4700
Participants
  Yes | 4539
  No | 161

ADVERSE EVENTS:
Time Frame: From start of treatment until end of observation or discontinuation of treatment, whichever occurred first, up to 29 weeks.
Description: Treated set (TS): All screened patients with informed consent, date of registration (date of creation of screening form in the Electronic Case Report Form (eCRF)), and at least one documented administration of Spiolto® Respimat®.
Arm/Group | Spiolto® Respimat®
All-Cause Mortality (participants affected / at risk) | 7/4819
Serious Adverse Events (participants affected / at risk) | 8/4819
Other Adverse Events (participants affected / at risk) | 0/4819
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spiolto® Respimat® (N=4819)
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Loss of consciousness (Nervous system disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Death (General disorders) | 3
Sudden death (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/69/NCT03663569/Prot_002.pdf
  • Statistical Analysis Plan (2019-07-19): https://cdn.clinicaltrials.gov/large-docs/69/NCT03663569/SAP_001.pdf